CLINICAL TRIAL: NCT02190838
Title: Phase II Multicenter Randomized Study to Compare Dacarbazine With Melatonin or Metformin Versus Dacarbazine in the First Line Therapy of Disseminated Melanoma
Brief Title: Comparison of Melatonin or Metformin and Dacarbazine Combination Versus Dacarbazine Alone in Disseminated Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Preliminary terminated due to inefficacy
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMM-1
Record Dates: First submitted 2014-07-13; First posted 2014-07-15 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-09

CONDITIONS: Melanoma
Keywords: Melanoma; Melatonin; Metformin; Dacarbazine
MeSH Terms: conditions — Melanoma | interventions — Metformin; Melatonin; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dacarbazine with Metformin (Experimental): 32 patients will receive Dacarbazine 1000 mg/m^2 once every 28 days with Metformin 850 mg BID.
  Interventions: Drug: Metformin; Drug: Dacarbazine
- Dacarbazine and Melatonin (Experimental): 32 patients will receive Dacarbazine 1000 mg/m^2 once every 28 days with Melatonin 3 mg before sleep daily.
  Interventions: Drug: Melatonin; Drug: Dacarbazine
- Dacarbazine (Active Comparator): 32 patients will receive Dacarbazine 1000 mg/m^2 once every 28 days
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: Metformin — per os 850 mg BID
  Other Names: Siofor® 850
  Arms: Dacarbazine with Metformin
Drug: Melatonin — per os 3 mg daily
  Other Names: Melaxen
  Arms: Dacarbazine and Melatonin
Drug: Dacarbazine — IV 1 hour 1000 mg/m^2 once in 28 days
  Other Names: DTIC

SUMMARY:
Treatment of disseminated melanoma is still a difficult issue. Obvious achievements of recent years proves efficacy of immunologic approachees in this field. The ability of melatonin and metformin to decrease metabolic immunosuppression was shown in many experimental studies. Some literature data confirm the possibility of increasing efficacy of melatonin with dacarbazine (DTIC) and metformin with DTIC combinations. We hypothesized that this combinations could be more effective than DTIC monotherapy in terms of response rate and time to progression.

ELIGIBILITY:
Inclusion Criteria:

* Age >18.
* Obtained Inform Consent
* Morphologically confirmed disseminated Stage IV melanoma
* Eastern Collaborative Oncology Group Performance Status Scale 0 - 2.
* Expected survival >3 month

Exclusion Criteria:

* Evidence of active brain lesions (brain lesions after stereotaxic ray therapy allowed)
* Evidence of liver and bone marrow clinically meaningful disfunction
* Severe uncontrolled concomitant conditions and diseases
* Pregnancy or lactation
* Systemic therapy for disseminated melanoma
* Second malignancy
* Diabetes mellitus requiring drug therapy
* Any condition preventing study participation by investigator opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-12-12 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Response Rate | 23 months after FPFV
  Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. ORR is defined as the proportion of patients with a best overall response of complete response or partial response
Progression Free Survival | 23 months after FPFV
  As per RECIST v1.1. progression-free survival (PFS) is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause.

SECONDARY OUTCOMES:
Adverse events (AE) incidence | until 30 days after last patient treatment visit
  Incidence of AE classified using NCI Common Terminology Criteria for AE v4
Metabolic Changes Incidence | 23 months after FPFV
  Nutritional status will be assessed using Nutritional Risk Index (NRI), Subjective global assessment (SGA), and Body Mass Index (BMI) tools.
Immune system assessment | 23 months after FPFV
  Following tests will be performed at baseline and each response assessment:
  * Lymphocyte subpopulations detection
  * Immunosuppressive factors measurements

CONTACTS AND LOCATIONS:
Overall Officials: Aleksei V. Novik, MD, PhD, Principal Investigator — N.N. Petrov Research Institute of Oncology; Irina A. Baldueva, MD, PhD, DSc, Study Director — N.N. Petrov Research Institute of Oncology
Locations (3):
- Russia (3):
  - N.N. Petrov Research Institute of Oncology Clinical Diagnostic Department, Saint Petersburg
  - N.N. Petrov Research Institute of Oncology Ambulatory Chemotherapy Department, Saint Petersburg
  - N.N. Petrov Research Institute of Oncology Chemotherapy and Innovative Technologies Department, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Novik AV, Protsenko SA, Baldueva IA, Berstein LM, Anisimov VN, Zhuk IN, Semenova AI, Latipova DK, Tkachenko EV, Semiglazova TY. Melatonin and Metformin Failed to Modify the Effect of Dacarbazine in Melanoma. Oncologist. 2021 May;26(5):364-e734. doi: 10.1002/onco.13761. Epub 2021 Apr 9. PMID 33749049